CLINICAL TRIAL: NCT01496105
Title: Efficacy Study of Topical Application of Lidacaine Spray Prior to IUD Insertion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Saied Eldin Elsafty, Lecturer of Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ali elyan 2011
Record Dates: First submitted 2011-12-13; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Drug Usage
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocaine spray 10% (Active Comparator)
  Interventions: Drug: Lidocaine
- Saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Lidocaine
  Arms: lidocaine spray 10%
Drug: saline
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether the topical use of lidocaine spray 10% on the cervix is an effective way to reduce pain during IUCD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Speak Arabic or English

Exclusion Criteria:

* History of cervical surgery
* Known hypersensitivity to topical analgesics
* First trimester abortion or miscarriage in the previous six weeks
* Second trimester abortion or miscarriage in the previous 12 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
VAS score of Pain | 5 minutes from lidocaine spraying ( after application of tenaculum)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospital, Cairo, Egypt